CLINICAL TRIAL: NCT05985369
Title: The Effects of a High-quality Vegan Diet on Skeletal Muscle Maintenance and Adaptation in Comparison to a Protein-matched Omnivorous Diet in Healthy Older Adults.
Brief Title: Vegan and Omnivorous Diets and Skeletal Muscle Turnover in Healthy Older Adults
Acronym: MVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 524790
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy Aging
Keywords: Muscle metabolism; Protein metabolism; Sarcopenia; Resistance exercise
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegan diet (Experimental): Participants will be allocated to a fully controlled 1-week vegan diet containing 0.8 g/kg BW/day of protein where all protein provided will be derived from non-animal-derived protein sources.
  Interventions: Other: Controlled diet and resistance exercise
- Omnivorous diet (Experimental): Participants will be allocated to a fully controlled 1-week omnivorous diet containing 0.8 g/kg BW/day of protein where the majority of protein will be derived from animal-derived protein sources.
  Interventions: Other: Controlled diet and resistance exercise

INTERVENTIONS:
Other: Controlled diet and resistance exercise — Participants will adopt a 1-week completely controlled diet and perform 3 sessions of unilateral leg resistance exercise.

SUMMARY:
Dietary protein intake and physical activity are key to minimise the age-related loss of skeletal muscle mass. While animal-derived protein sources are considered high-quality anabolic foods, it remains unclear whether non-animal-derived (vegan) protein sources support skeletal muscle maintenance and healthy ageing. The aim of the present study is to assess the effect of a vegan diet on daily muscle protein synthesis rates compared to a protein-matched omnivorous diet where the majority of protein is derived from high-quality animal-based protein sources.

DETAILED DESCRIPTION:
Background: The age-related loss of muscle mass and strength is (partly) explained by a blunted responsiveness of skeletal muscle to the anabolic properties of dietary protein and muscle contraction. Therefore, sufficient dietary protein intake and physical activity are required to minimise age-related muscle atrophy. It remains unknown whether this can be achieved utilising non-animal-derived (vegan) protein sources.

Objective: To assess daily muscle protein synthesis rates when adopting a vegan or protein-matched omnivorous control diet.

Methods: Healthy older adults (aged 60-80 years) will be randomly allocated to a completely controlled 1-week vegan (providing 0.8 g/kg BW/day protein) or protein-matched omnivorous diet. During this week, participants will perform a set of unilateral leg resistance exercise on day 1, 3, and 5. Deuterium oxide in combination with saliva and muscle sample (from the m. vastus lateralis) collection will be used to measure daily muscle protein synthesis rates in resting and exercised tissue.

Value: This will be the first study assessing daily muscle protein turnover in healthy older adults adopting a 1-week vegan diet. This will contribute to the understanding and viability of vegan protein to support active and healthy ageing.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 - 30
* Active (not very sedentary and not master athlete; assessed via IPAQ)
* Women only: post menopause

Exclusion Criteria:

* Hypertension (>150/90 mmHg)
* Any diagnosed metabolic impairment
* Any diagnosed cardiovascular disease
* Any diagnosed gastrointestinal disease
* Diagnosed cancer
* Any medication known to affect muscle metabolism (e.g. hormone replacement therapy)
* Severe food allergies or intolerances (e.g. celiac, lactose intolerance, allergic to fungi or algae foods)
* Smoking

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis (MPS) in resting and exercised tissue | 7 days
  Daily MPS rates, expressed as fractional synthetic rate (%/h)

SECONDARY OUTCOMES:
Muscle morphology | 7 days
  Changes in muscle thickness during the intervention period, measured via ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, Devond, United Kingdom